CLINICAL TRIAL: NCT02276521
Title: Evaluation of Long-term Immunological Responses Following Reduced Dose Quadrivalent Human Papillomavirus (HPV) Vaccine Schedules: A Phase II/III Clinical Trial
Brief Title: Evaluation of Long Term Immunity Following HPV Vaccination
Status: Completed | Type: Observational
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Department of Foregin Affairs and Trade, Australia (Other Government); Ministry of Health, Fiji (Other Government); The Royal Women Hospital (Unknown); Colonial War Memorial Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2014.5.FNRERC.5.SU
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Cervical Cancer; Anogenital Warts
MeSH Terms: conditions — Uterine Cervical Neoplasms; Condylomata Acuminata | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — We will be collecting blood from the participants, which include the plasma and peripheral blood mononuclear cells.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Zero dose group: Participants that did not received any HPV vaccine previously.
  Interventions: Biological: Cervarix®
- One dose group: Participants that received one dose of Gardasil® vaccine 5-6 years ago from a vaccination campaign.
  Interventions: Biological: Cervarix®
- Two dose group: Participants that received two dose of Gardasil® vaccine 5-6 years ago from a vaccination campaign.
  Interventions: Biological: Cervarix®
- Three dose group: Participants that received three dose of Gardasil® vaccine 5-6 years ago from a vaccination campaign.
  Interventions: Biological: Cervarix®

INTERVENTIONS:
Biological: Cervarix® — All groups will received one dose of Cervarix® vaccine

SUMMARY:
In Fiji, cervical cancer is the second most frequent cancer and the highest cause of cancer mortality in women. In 2008/9, the Ministry of Health in Fiji accepted a donation of 110,000 doses of quadrivalent HPV vaccine, Gardasil® based on the high cervical cancer disease burden. There was enough vaccine to vaccinate all girls aged 9-12 years (30,338 girls) with a three-dose schedule, but not all girls received three doses of the vaccine. This means those girls that received reduced doses may not be fully protected against the HPV genotypes present in the Gardasil®. While HPV vaccines are highly immunogenic and efficacious in the licensed three-dose schedule, there is limited information about the effectiveness of reduced dose schedules in terms of immunogenicity and memory. There is growing evidence from other studies that two doses of HPV vaccine may be sufficient for protection. Reduced schedules would be of benefit in Fiji due to improved costs and logistics. This study will examine whether one or two doses of HPV vaccine provide similar immunological evidence of long-term protection to the standard three-dose schedule in terms of antibody titres to the genotypes present in the Gardasil®. To compare immunological memory responses between dosage groups, a dose of Cervarix ® will be administered to all girls so that the magnitude of the memory responses can be measured.

DETAILED DESCRIPTION:
In 2008/9, the Ministry of Health (MoH) in Fiji accepted a donation of 110,000 doses of quadrivalent HPV vaccine, Gardasil® based on the high cervical cancer disease burden. There was enough vaccine to vaccinate all girls aged 9-12 years (30,338 girls) with a three-dose schedule, but not all girls received three doses of the vaccine. This means those girls that received reduced doses may not be fully protected against the HPV genotypes present in the Gardasil®. In 2013, the Fiji MoH with Australian Aid support introduced the Cervarix ® vaccine as a three dose schedule (0, 1, and 6 months) to be given to all girls at the last year of primary school as part of the national immunisation program. This is a unique opportunity to determine if fewer than three doses of Gardasil® vaccine are immunologically similar to the standard three-dose schedule 6 years after receiving the vaccine (ie indicating long-term protection).

This is an open label Phase II/III clinical trial in girls (now aged 14-17 years) who previously received zero, one, two or three doses of Gardasil® in 2008/9. A dose of Cervarix ® will be administered to all the girls in this study so that immunological evidence of long-term protection in terms of antibody levels (including neutralisation titres), number of memory B and T cells (including cytokine responses) and gene expression profiles can be measured.

A non-random sample of 200 girls will be recruited; girls previously received one, two or three doses of Gardasil® will be identified through school vaccination lists obtained from the MoH and Ministry of Education; girls that did not receive any vaccines previously will be recruited via recommendations of friends of the girls and by informal networks. The investigators aim to have approximately 50% indigenous Fijian (i-Taukei)/others and 50% Fijians of Indian descent in the study.

Informed consents will be obtained from both the parent/guardian of the participant and the participant, as well as checking the participant's eligibility by the study nurses. Twenty-five milliliters (mL) of blood in total will be drawn from each participant before and 28 days after a dose of Cervarix® vaccine. To ensure all participants receive three doses of HPV vaccine by the end of study, follow up appointments will be made for study participants to receive off-study vaccine for those that did not receive any HPV vaccine previously or received only one dose of Gardasil® in 2008/9 campaign; no samples will be collected in the follow-up appointments.

Peripheral blood mononuclear cells (PBMC) and plasma will be separated from the blood, and freeze down down in liquid nitrogen and -80 degree freezer until laboratory analysis, respectively.

Sample size:

The primary outcome is the comparison of the geometric mean concentrations (GMCs) of HPV- specific antibody responses (including neutralisation titres) against HPV 6, -11, -16 and -18, between the groups that previously received zero, one, two or three doses of Gardasil®. Based on published data from a 5 year follow-up study (Olsson et al. 2007), the standard deviations for anti-HPV antibodies are 570 (HPV16) and 84 (HPV18). The sample size required to provide 80% power to detect a 30% difference in HPV antibodies ranges from 48/group (HPV16) to 49/group (HPV18). A sample size of 50/group will be used in this study.

Statistical Analysis Plan:

Comparison of GMCs of anti-HPV antibody levels and neutralising antibody levels will be compared using log-transformed data using the Student's t-test. The proportion with seropositivity will be compared using the Fisher's exact test. These analyses will also be used to compare anti-HPV antibody levels and neutralising antibody levels one month post Cervarix®. Comparison of B- and T- cell frequencies will be done using the Mann-Whitney U test. For cytokine secretion in PBMC supernatants, comparison of GMCs ± 95% confidence intervals (CI) will be done on log-transformed data using the Student's t-test. The gene expression profiles (tumour necrosis factor-α, interleukin (IL)- 6, IL-8, interferon-γ, IL-18 and IL-1β) in different groups will be compared using a paired student t test. The fold increase or decrease in the gene expression will be assessed using the sign test. A p-value <0.05 will be considered statistically significant for all analyses.

Data Collection:

Each child will have a unique study number and folder collating the field site study case report forms (CRFs). All laboratory processing will be undertaken in a blinded fashion using de-identified samples. Field and clinical data will be entered in the study office by trained study staff using the EpiData software and sent to Drs Russell and Licciardi for analysis. The design of the computer databases and data cleaning will be done by the study staff under supervision of the principal investigators. Only designated study staff and the investigators associated with this project will have access to this data. Data will be analysed with help of staff from Clinical Epidemiology and Biostatistics Unit (CEBU), Murdoch Childrens Research Institute (MCRI).

Data Storage:

All laboratory data collected in this study will be stored electronically and in hard copy format and secured in lockable filing cabinets for 15 years after the completion of the study.

Study Record Retention:

The biological samples will be stored at the Immunology Laboratory at MCRI for 15 years following completion of the study, in accordance to ethics requirements for a clinical trial. The samples will be destroyed if the participants do not consent for their blood sample to be used for further ethics approved HPV related studies. If the participant consent for their blood sample to be used for future ethically approved research, related to this study only, the samples will be kept indefinitely at MCRI, Melbourne, Australia. Additional ethics approval is required if the investigators wish to use these future use samples later on for HPV related studies.

All the consent forms will be filed in proper folders and secured in lockable filing cabinets on-site in Fiji for 15 years following completion of the study. The consent forms will be shredded and disposed in locked security bins.

All participating investigators and research staff will maintain subject confidentiality. Except for the consent form, participants will be identified only by their unique study number throughout the study. This extends to the clinical information, testing of the biological samples, documentation, and laboratory database.

Parents/guardians will be reimbursed for their time and travel for the sample collection.

MCRI and Fiji MoH have signed a Memorandum of Understanding (MoU). A Research Specific Agreement is being developed by the Fiji MoH and MCRI which will include intellectual property and publication clauses. The agreement to be developed will not unreasonably delay the publication of results from the study, or harm or prejudice an outcome of the research program or an interest a party has in intellectual property, either developed pursuant to the research program or that owned by the party.

ELIGIBILITY:
Inclusion Criteria:

* Girls who live in Suva and were previously vaccinated with one, two or three Gardasil® doses or were eligible but did not receive Gardasil® vaccine in the 2008/9 campaign will be eligible for the study.

Exclusion Criteria:

* Any participant who had anaphylaxis following a previous dose of the vaccine, anaphylaxis to any vaccine component, or possible pregnancy will be excluded from this study.
* In addition, any participant whose dates of previous Gardasil® vaccination are uncertain, or has received Cervarix® vaccine previously, or has an axillary temperature greater than 38°C will be excluded from this study.

Ages: 15 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In 2008/9, the MoH in Fiji accepted a one-off donation of 110,000 doses of Gardasil® vaccine, which was enough to vaccinate four birth cohorts of girls (30,338 girls aged 9-12 years) with a three-dose schedule via a school-based program. However, not all the girls received the full-recommended three-dose schedule, mainly due to absence from school on the day the school health team were visiting. The coverage following the initial and the subsequent mop-up campaign was: 62%, 56%, and 55% for doses one, two, and three respectively. The girls that received different doses of Gardasil® vaccine in Suva area who are potentially contactable in this study are 676 (three doses), 204 (two doses) and 116 (one dose), demonstrating feasibility of recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
GMCs of HPV- specific antibody titres against HPV 6, 11, 16 and 18 | 6 months

SECONDARY OUTCOMES:
GMCs of HPV- specific antibody titres against HPV 6, 11, 16 and 18 one month post Cervarix® | 6 months
Number of HPV- specific memory B- and T- cells against HPV 6, 11, 16 and 18 pre and one month post Cervarix® | 11 months
Fold change in the gene expression profiles in immune cells both pre- and one month post Cervarix® | 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward K Mulholland, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Colonial War Memorial Hospital, Suva, Fiji

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] de Sanjose S, Quint WG, Alemany L, Geraets DT, Klaustermeier JE, Lloveras B, Tous S, Felix A, Bravo LE, Shin HR, Vallejos CS, de Ruiz PA, Lima MA, Guimera N, Clavero O, Alejo M, Llombart-Bosch A, Cheng-Yang C, Tatti SA, Kasamatsu E, Iljazovic E, Odida M, Prado R, Seoud M, Grce M, Usubutun A, Jain A, Suarez GA, Lombardi LE, Banjo A, Menendez C, Domingo EJ, Velasco J, Nessa A, Chichareon SC, Qiao YL, Lerma E, Garland SM, Sasagawa T, Ferrera A, Hammouda D, Mariani L, Pelayo A, Steiner I, Oliva E, Meijer CJ, Al-Jassar WF, Cruz E, Wright TC, Puras A, Llave CL, Tzardi M, Agorastos T, Garcia-Barriola V, Clavel C, Ordi J, Andujar M, Castellsague X, Sanchez GI, Nowakowski AM, Bornstein J, Munoz N, Bosch FX; Retrospective International Survey and HPV Time Trends Study Group. Human papillomavirus genotype attribution in invasive cervical cancer: a retrospective cross-sectional worldwide study. Lancet Oncol. 2010 Nov;11(11):1048-56. doi: 10.1016/S1470-2045(10)70230-8. Epub 2010 Oct 15. PMID 20952254
- [Background] Winer RL, Kiviat NB, Hughes JP, Adam DE, Lee SK, Kuypers JM, Koutsky LA. Development and duration of human papillomavirus lesions, after initial infection. J Infect Dis. 2005 Mar 1;191(5):731-8. doi: 10.1086/427557. Epub 2005 Jan 21. PMID 15688287
- [Background] Teissier S, Pang CL, Thierry F. The E2F5 repressor is an activator of E6/E7 transcription and of the S-phase entry in HPV18-associated cells. Oncogene. 2010 Sep 9;29(36):5061-70. doi: 10.1038/onc.2010.246. Epub 2010 Jul 19. PMID 20639900
- [Background] Sellors JW, Karwalajtys TL, Kaczorowski J, Mahony JB, Lytwyn A, Chong S, Sparrow J, Lorincz A; Survey of HPV in Ontario Women Group. Incidence, clearance and predictors of human papillomavirus infection in women. CMAJ. 2003 Feb 18;168(4):421-5. PMID 12591782
- [Background] Kanodia S, Fahey LM, Kast WM. Mechanisms used by human papillomaviruses to escape the host immune response. Curr Cancer Drug Targets. 2007 Feb;7(1):79-89. doi: 10.2174/156800907780006869. PMID 17305480
- [Background] Stanley M. Immune responses to human papillomavirus. Vaccine. 2006 Mar 30;24 Suppl 1:S16-22. doi: 10.1016/j.vaccine.2005.09.002. PMID 16219398
- [Background] Kirnbauer R, Hubbert NL, Wheeler CM, Becker TM, Lowy DR, Schiller JT. A virus-like particle enzyme-linked immunosorbent assay detects serum antibodies in a majority of women infected with human papillomavirus type 16. J Natl Cancer Inst. 1994 Apr 6;86(7):494-9. doi: 10.1093/jnci/86.7.494. PMID 8133532
- [Background] Who. Human papillomavirus vaccines: WHO position paper. Biologicals. 2009 Oct;37(5):338-44. doi: 10.1016/j.biologicals.2009.04.005. Epub 2009 Jun 13. No abstract available. PMID 19525124
- [Background] Garcon N, Wettendorff M, Van Mechelen M. Role of AS04 in human papillomavirus vaccine: mode of action and clinical profile. Expert Opin Biol Ther. 2011 May;11(5):667-77. doi: 10.1517/14712598.2011.573624. Epub 2011 Apr 4. PMID 21457083
- [Background] Joura EA, Leodolter S, Hernandez-Avila M, Wheeler CM, Perez G, Koutsky LA, Garland SM, Harper DM, Tang GW, Ferris DG, Steben M, Jones RW, Bryan J, Taddeo FJ, Bautista OM, Esser MT, Sings HL, Nelson M, Boslego JW, Sattler C, Barr E, Paavonen J. Efficacy of a quadrivalent prophylactic human papillomavirus (types 6, 11, 16, and 18) L1 virus-like-particle vaccine against high-grade vulval and vaginal lesions: a combined analysis of three randomised clinical trials. Lancet. 2007 May 19;369(9574):1693-702. doi: 10.1016/S0140-6736(07)60777-6. PMID 17512854
- [Background] FUTURE II Study Group. Quadrivalent vaccine against human papillomavirus to prevent high-grade cervical lesions. N Engl J Med. 2007 May 10;356(19):1915-27. doi: 10.1056/NEJMoa061741. PMID 17494925
- [Background] Harper DM, Franco EL, Wheeler C, Ferris DG, Jenkins D, Schuind A, Zahaf T, Innis B, Naud P, De Carvalho NS, Roteli-Martins CM, Teixeira J, Blatter MM, Korn AP, Quint W, Dubin G; GlaxoSmithKline HPV Vaccine Study Group. Efficacy of a bivalent L1 virus-like particle vaccine in prevention of infection with human papillomavirus types 16 and 18 in young women: a randomised controlled trial. Lancet. 2004 Nov 13-19;364(9447):1757-65. doi: 10.1016/S0140-6736(04)17398-4. PMID 15541448
- [Background] Villa LL, Costa RL, Petta CA, Andrade RP, Paavonen J, Iversen OE, Olsson SE, Hoye J, Steinwall M, Riis-Johannessen G, Andersson-Ellstrom A, Elfgren K, Krogh Gv, Lehtinen M, Malm C, Tamms GM, Giacoletti K, Lupinacci L, Railkar R, Taddeo FJ, Bryan J, Esser MT, Sings HL, Saah AJ, Barr E. High sustained efficacy of a prophylactic quadrivalent human papillomavirus types 6/11/16/18 L1 virus-like particle vaccine through 5 years of follow-up. Br J Cancer. 2006 Dec 4;95(11):1459-66. doi: 10.1038/sj.bjc.6603469. Epub 2006 Nov 21. PMID 17117182
- [Background] Villa LL, Ault KA, Giuliano AR, Costa RL, Petta CA, Andrade RP, Brown DR, Ferenczy A, Harper DM, Koutsky LA, Kurman RJ, Lehtinen M, Malm C, Olsson SE, Ronnett BM, Skjeldestad FE, Steinwall M, Stoler MH, Wheeler CM, Taddeo FJ, Yu J, Lupinacci L, Railkar R, Marchese R, Esser MT, Bryan J, Jansen KU, Sings HL, Tamms GM, Saah AJ, Barr E. Immunologic responses following administration of a vaccine targeting human papillomavirus Types 6, 11, 16, and 18. Vaccine. 2006 Jul 7;24(27-28):5571-83. doi: 10.1016/j.vaccine.2006.04.068. Epub 2006 May 15. PMID 16753240
- [Background] Giannini SL, Hanon E, Moris P, Van Mechelen M, Morel S, Dessy F, Fourneau MA, Colau B, Suzich J, Losonksy G, Martin MT, Dubin G, Wettendorff MA. Enhanced humoral and memory B cellular immunity using HPV16/18 L1 VLP vaccine formulated with the MPL/aluminium salt combination (AS04) compared to aluminium salt only. Vaccine. 2006 Aug 14;24(33-34):5937-49. doi: 10.1016/j.vaccine.2006.06.005. Epub 2006 Jun 19. PMID 16828940
- [Background] Harper DM, Franco EL, Wheeler CM, Moscicki AB, Romanowski B, Roteli-Martins CM, Jenkins D, Schuind A, Costa Clemens SA, Dubin G; HPV Vaccine Study group. Sustained efficacy up to 4.5 years of a bivalent L1 virus-like particle vaccine against human papillomavirus types 16 and 18: follow-up from a randomised control trial. Lancet. 2006 Apr 15;367(9518):1247-55. doi: 10.1016/S0140-6736(06)68439-0. PMID 16631880
- [Background] Rowhani-Rahbar A, Alvarez FB, Bryan JT, Hughes JP, Hawes SE, Weiss NS, Koutsky LA. Evidence of immune memory 8.5 years following administration of a prophylactic human papillomavirus type 16 vaccine. J Clin Virol. 2012 Mar;53(3):239-43. doi: 10.1016/j.jcv.2011.12.009. Epub 2011 Dec 30. PMID 22209292
- [Background] Villa LL, Costa RL, Petta CA, Andrade RP, Ault KA, Giuliano AR, Wheeler CM, Koutsky LA, Malm C, Lehtinen M, Skjeldestad FE, Olsson SE, Steinwall M, Brown DR, Kurman RJ, Ronnett BM, Stoler MH, Ferenczy A, Harper DM, Tamms GM, Yu J, Lupinacci L, Railkar R, Taddeo FJ, Jansen KU, Esser MT, Sings HL, Saah AJ, Barr E. Prophylactic quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in young women: a randomised double-blind placebo-controlled multicentre phase II efficacy trial. Lancet Oncol. 2005 May;6(5):271-8. doi: 10.1016/S1470-2045(05)70101-7. PMID 15863374
- [Background] Wrammert J, Ahmed R. Maintenance of serological memory. Biol Chem. 2008 May;389(5):537-9. doi: 10.1515/bc.2008.066. PMID 18953719
- [Background] Ohlschlager P, Osen W, Dell K, Faath S, Garcea RL, Jochmus I, Muller M, Pawlita M, Schafer K, Sehr P, Staib C, Sutter G, Gissmann L. Human papillomavirus type 16 L1 capsomeres induce L1-specific cytotoxic T lymphocytes and tumor regression in C57BL/6 mice. J Virol. 2003 Apr;77(8):4635-45. doi: 10.1128/jvi.77.8.4635-4645.2003. PMID 12663770
- [Background] Mariani L, Venuti A. HPV vaccine: an overview of immune response, clinical protection, and new approaches for the future. J Transl Med. 2010 Oct 27;8:105. doi: 10.1186/1479-5876-8-105. PMID 20979636
- [Background] Kreimer AR, Rodriguez AC, Hildesheim A, Herrero R, Porras C, Schiffman M, Gonzalez P, Solomon D, Jimenez S, Schiller JT, Lowy DR, Quint W, Sherman ME, Schussler J, Wacholder S; CVT Vaccine Group. Proof-of-principle evaluation of the efficacy of fewer than three doses of a bivalent HPV16/18 vaccine. J Natl Cancer Inst. 2011 Oct 5;103(19):1444-51. doi: 10.1093/jnci/djr319. Epub 2011 Sep 9. PMID 21908768
- [Background] Romanowski B, Schwarz TF, Ferguson LM, Peters K, Dionne M, Schulze K, Ramjattan B, Hillemanns P, Catteau G, Dobbelaere K, Schuind A, Descamps D. Immunogenicity and safety of the HPV-16/18 AS04-adjuvanted vaccine administered as a 2-dose schedule compared with the licensed 3-dose schedule: results from a randomized study. Hum Vaccin. 2011 Dec;7(12):1374-86. doi: 10.4161/hv.7.12.18322. Epub 2011 Dec 1. PMID 22048171
- [Background] Dobson SR, McNeil S, Dionne M, Dawar M, Ogilvie G, Krajden M, Sauvageau C, Scheifele DW, Kollmann TR, Halperin SA, Langley JM, Bettinger JA, Singer J, Money D, Miller D, Naus M, Marra F, Young E. Immunogenicity of 2 doses of HPV vaccine in younger adolescents vs 3 doses in young women: a randomized clinical trial. JAMA. 2013 May 1;309(17):1793-802. doi: 10.1001/jama.2013.1625. PMID 23632723
- [Background] Olsson SE, Villa LL, Costa RL, Petta CA, Andrade RP, Malm C, Iversen OE, Hoye J, Steinwall M, Riis-Johannessen G, Andersson-Ellstrom A, Elfgren K, von Krogh G, Lehtinen M, Paavonen J, Tamms GM, Giacoletti K, Lupinacci L, Esser MT, Vuocolo SC, Saah AJ, Barr E. Induction of immune memory following administration of a prophylactic quadrivalent human papillomavirus (HPV) types 6/11/16/18 L1 virus-like particle (VLP) vaccine. Vaccine. 2007 Jun 21;25(26):4931-9. doi: 10.1016/j.vaccine.2007.03.049. Epub 2007 Apr 20. PMID 17499406
- [Background] Smolen KK, Gelinas L, Franzen L, Dobson S, Dawar M, Ogilvie G, Krajden M, Fortuno ES 3rd, Kollmann TR. Age of recipient and number of doses differentially impact human B and T cell immune memory responses to HPV vaccination. Vaccine. 2012 May 21;30(24):3572-9. doi: 10.1016/j.vaccine.2012.03.051. Epub 2012 Mar 31. PMID 22469863
- [Background] Dauner JG, Pan Y, Hildesheim A, Harro C, Pinto LA. Characterization of the HPV-specific memory B cell and systemic antibody responses in women receiving an unadjuvanted HPV16 L1 VLP vaccine. Vaccine. 2010 Jul 26;28(33):5407-13. doi: 10.1016/j.vaccine.2010.06.018. Epub 2010 Jun 17. PMID 20591543
- [Background] Law I, Fong JJ, Buadromo EM, Samuela J, Patel MS, Garland SM, Mulholland EK, Russell FM. The high burden of cervical cancer in Fiji, 2004-07. Sex Health. 2013 May;10(2):171-8. doi: 10.1071/SH12135. PMID 23557630
- [Background] Tabrizi SN, Law I, Buadromo E, Stevens MP, Fong J, Samuela J, Patel M, Mulholland EK, Russell FM, Garland SM. Human papillomavirus genotype prevalence in cervical biopsies from women diagnosed with cervical intraepithelial neoplasia or cervical cancer in Fiji. Sex Health. 2011 Sep;8(3):338-42. doi: 10.1071/SH10083. PMID 21851773
- [Background] Neuzil KM, Canh DG, Thiem VD, Janmohamed A, Huong VM, Tang Y, Diep NT, Tsu V, LaMontagne DS. Immunogenicity and reactogenicity of alternative schedules of HPV vaccine in Vietnam: a cluster randomized noninferiority trial. JAMA. 2011 Apr 13;305(14):1424-31. doi: 10.1001/jama.2011.407. PMID 21486975
- [Background] Centers for Disease Control and Prevention (CDC). FDA licensure of bivalent human papillomavirus vaccine (HPV2, Cervarix) for use in females and updated HPV vaccination recommendations from the Advisory Committee on Immunization Practices (ACIP). MMWR Morb Mortal Wkly Rep. 2010 May 28;59(20):626-9. PMID 20508593
- [Background] Descamps D, Hardt K, Spiessens B, Izurieta P, Verstraeten T, Breuer T, Dubin G. Safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine for cervical cancer prevention: a pooled analysis of 11 clinical trials. Hum Vaccin. 2009 May;5(5):332-40. doi: 10.4161/hv.5.5.7211. Epub 2009 May 20. PMID 19221517
- [Background] Gold MS, McIntyre P. Human papillomavirus vaccine safety in Australia: experience to date and issues for surveillance. Sex Health. 2010 Sep;7(3):320-4. doi: 10.1071/SH09153. PMID 20719221
- [Background] Tabrizi SN, Frazer IH, Garland SM. Serologic response to human papillomavirus 16 among Australian women with high-grade cervical intraepithelial neoplasia. Int J Gynecol Cancer. 2006 May-Jun;16(3):1032-5. doi: 10.1111/j.1525-1438.2006.00587.x. PMID 16803481